CLINICAL TRIAL: NCT04450329
Title: A Phase III Randomised, Double-masked, Parallel Group, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity Between SB15 (Proposed Aflibercept Biosimilar) and Eylea® in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: A Study to Compare SB15 (Proposed Aflibercept Biosimilar) to Eylea in Subjects With Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB15-3001
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SB15 (Proposed aflibercept biosimilar) (Experimental): Subjects randomized into SB15 group will receive SB15 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
  Interventions: Drug: SB15 (Proposed aflibercept biosimilar)
- Eylea (Aflibercept) (Active Comparator): Subjects randomized into Eylea group will receive Eylea 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
  At Week 32, subjects in Eylea group will re-randomized into SB15 or Eylea group. After re-randomization, subjects transited to SB15 group will receive SB15 2 mg (0.05 mL) once every 8 weeks until Week 48 and subjects remaining in Eylea group will continue to receive Eylea 2 mg (0.05 mL) once every 8 weeks until Week 48.
  Interventions: Drug: SB15 (Proposed aflibercept biosimilar); Drug: Eylea (Aflibercept)

INTERVENTIONS:
Drug: SB15 (Proposed aflibercept biosimilar) — Subjects randomized into SB15 group will receive SB15 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48. Starting at Week 32, subjects transited from Eylea to SB15 will receive SB15 2 mg (0.05 mL) via intravitreal injection every 8 weeks.
Drug: Eylea (Aflibercept) — Subjects randomized into Eylea group will receive Eylea 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
  Arms: Eylea (Aflibercept)

SUMMARY:
This is a randomised, double-masked, parallel group, multicentre study to evaluate the efficacy, safety, Pharmacokinetics (PK), and immunogenicity of SB15 compared to Eylea® in subjects with neovascular AMD.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either SB15 or Eylea® (administered via intravitreal [IVT] injection 2 mg [0.05 mL] every 4 weeks for the first 3 months (i.e., at Weeks 0, 4, and 8), followed by 2 mg [0.05 mL] once every 8 weeks). At Week 32, subjects in Eylea® treatment group will be randomised again in a 1:1 ratio to either continue on Eylea® treatment or be transitioned to SB15 treatment. In the 8-week treatment cycle, IPs (SB15 or Eylea®) will be administered up to Week 48, and the last assessment will be done at Week 56, corresponding to the end of follow-up for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years at Screening
2. Treatment naïve, *active subfoveal choroidal neovascularisation (CNV) lesion secondary to AMD in the study eye
3. The area of CNV must occupy at least 50% of total lesion in the study eye
4. Total lesion area ≤ 9.0 Disc Areas (DA) in size (including blood, scars, and neovascularisation) in the study eye
5. BCVA of 20/40 to 20/200 (letter score of 73 to 34, inclusive) using ETDRS charts or 2702 series Number charts in the study eye at Screening and at Week 0 (Day 1) prior to randomisation
6. Non-childbearing potential female, OR childbearing potential female subjects or male subjects with their (respectively male or female) partners who agree to use at least two forms of appropriate contraception method that can achieve a failure rate of less than 1% per year from Screening until 3 months after the last IVT injection of IP
7. Written informed consent form (ICF) must be obtained from the subject prior to any study related procedure
8. Willingness and ability to undertake all scheduled visits and assessments

Exclusion Criteria:

1. Study eye: Sub- or intra-retinal haemorrhage that comprises more than 50% of the entire lesion or presence of blood with the size of 1 DA or more involving the centre of fovea
2. Study eye: Scar, fibrosis, or atrophy involving the centre of the fovea
3. Study eye: Presence of CNV due to other causes, such as ocular histoplasmosis, trauma, multifocal choroiditis, angioid streaks, history of choroidal rupture, or pathologic myopia
4. Study eye: Presence of retinal pigment epithelial tears or rips involving the macula
5. Study eye: Presence of macular hole at any stage
6. Study eye: Any concurrent macular abnormality other than AMD which could affect central vision or the efficacy of IP
7. Study eye: Any concurrent ocular condition which, in the opinion of the Investigator, could either confound the interpretation of efficacy and safety of IP or require medical or surgical intervention during the study period
8. Either eye: History or clinical evidence of diabetic retinopathy (except for mild non-proliferative diabetic retinopathy) or diabetic macular oedema (DME)
9. Study eye: Current vitreous haemorrhage
10. Either eye: Any previous IVT anti-vascular endothelial growth factor (VEGF) treatment
11. Any previous systemic anti-VEGF treatment
12. Study eye: History of treatment involving macula such as macular laser photocoagulation, photodynamic therapy (PDT), transpupillary thermotherapy (TTT), radiation therapy, or any ocular treatment for neovascular AMD
13. Any systemic treatment or therapy (including prescribed herbal medication) to treat neovascular AMD within 30 days prior to randomisation. However, dietary supplements, vitamins, or minerals will be allowed.
14. Study eye: History of vitrectomy, scleral buckling (encircling), glaucoma filtration surgery, corneal transplantation, or pan-retinal photocoagulation
15. Study eye: Previous ocular (intraocular and peribulbar) corticosteroids injection/implant within 1 year prior to randomisation
16. Study eye: Topical ocular corticosteroids administered for ≥ 30 consecutive days or for ≥ 60 nonconsecutive days within 90 days prior to randomisation
17. Use of systemic corticosteroids for 30 or more consecutive days within 90 days prior to randomization (inhaled steroid is permitted).
18. Study eye: Any other intraocular surgery or periocular surgery within 90 days prior to randomisation, except for lid surgery, which may not have taken place within 30 days prior to randomisation.
19. Current use of medications known to be toxic to the lens, retina, or optic nerve at Screening.
20. Study eye: Previous radiation therapy near the region of the study eye
21. Previous participation in clinical studies with IP to treat neovascular AMD in either eye.
22. Previous participation in clinical studies with IP to treat disease other than neovascular AMD within 90 days prior to randomisation (excluding dietary supplementary, vitamins, and minerals).
23. Subject with only one functional eye (defined as BCVA of counting finger or less on the eye with worse vision)
24. Study eye: Spherical equivalent of the refractive error demonstrating more than 6 diopters of myopia. For subjects who have undergone previous refractive or cataract surgery in the study eye, the preoperative refractive error in the study eye cannot exceed 6 diopters of myopia.
25. Study eye: Aphakia or absence of the posterior capsule (unless it occurred as a result of a YAG laser posterior capsulotomy in association with prior posterior chamber IOL implantation)
26. Either eye: Active or suspected ocular and periocular infection at Screening or at randomisation
27. Either eye: Active intraocular inflammation including scleritis at Screening or at randomisation
28. Either eye: History of idiopathic or autoimmune-associated uveitis
29. Study eye: Uncontrolled ocular hypertension (defined as intraocular pressure [IOP] ≥ 25 mmHg despite treatment with anti-glaucoma medication) at Screening
30. Known allergic reactions and/or hypersensitivity to any component of Eylea or SB15
31. History of allergy to the fluorescein sodium for injection in angiography
32. History of a medical condition that would preclude scheduled study visits or safe use of IP in the opinion of the Investigator
33. Uncontrolled systemic disease including but not limited to uncontrolled diabetes mellitus (in the opinion of the Investigator), uncontrolled systemic hypertension (systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 100 mmHg on optimal medical regimen), or uncontrolled atrial fibrillation (resting heart rate ≥ 110 beats per minutes) at Screening
34. Stroke, transient ischaemic attacks, or myocardial infarction within 180 days prior to randomisation
35. History of recurrent significant infections and/or current treatment for systemic infection
36. Severe renal impairment with dialysis or a history of renal transplant
37. Malignancy (other than non-melanoma skin cancer) under treatment or with history of metastatic disease
38. Women of childbearing potential who are pregnant, planning to become pregnant, lactating, or not using adequate birth control, as specified in protocol. For women of childbearing potential, a serum pregnancy test must result negative at Screening.
39. Employees of investigational sites, individuals directly involved with the conduct of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Se Joon Woo, Principal Investigator — Seoul National University Bundang Hospital, South Korea
Locations (38):
- United States (3):
  - SB Investigative Site, Colorado Springs, Colorado
  - SB Investigative Site, Chevy Chase, Maryland
  - SB Investigative Site, Abilene, Texas
- Croatia (2):
  - SB Investigative Site, Osijek
  - SB Investigative Site, Rijeka
- Czechia (3):
  - SB Investigative Site, Brno
  - SB Investigative Site, Hradec Králové
  - SB Investigative Site, Prague
- Estonia (2):
  - SB Investigative Site, Kohtla-Järve
  - SB Investigative Site, Tallinn
- Hungary (5):
  - SB Investigative Site, Budapest
  - SB Investigative Site, Debrecen
  - SB Investigative Site, Pécs
  - SB Investigative Site, Szeged
  - SB Investigative Site, Zalaegerszeg
- Japan (8):
  - SB Investigative Site, Aichi
  - SB Investigative Site, Fukuoka
  - SB Investigative Site, Inashiki-gun
  - SB Investigative Site, Kagoshima
  - SB Investigative Site, Nagasaki
  - SB Investigative Site, Osaka
  - SB Investigative Site, Saitama
  - SB Investigative Site, Tokyo
- SB Investigative Site, Riga, Latvia
- Poland (5):
  - SB Investigative Site, Bydgoszcz
  - SB Investigative Site, Katowice
  - SB Investigative Site, Krakow
  - SB Investigative Site, Lodz
  - SB Investigative Site, Tarnów
- Russia (4):
  - SB Investigative Site, Kovrov
  - SB Investigative Site, Moscow
  - SB Investigative Site, Novosibirsk
  - SB Investigative Site, Saint Petersburg
- South Korea (5):
  - SB Investigative Site, Ansan
  - SB Investigative Site, Busan
  - SB Investigative Site, Daegu
  - SB Investigative Site, Seongnam
  - SB Investigative Site, Seoul

REFERENCES:
- [Derived] Woo SJ, Bradvica M, Vajas A, Sagong M, Ernest J, Studnicka J, Veith M, Wylegala E, Patel S, Yun C, Orski M, Astakhov S, Toth-Molnar E, Csutak A, Enyedi L, Kim T, Oh I, Jang H, Sadda SR. Efficacy and Safety of the Aflibercept Biosimilar SB15 in Neovascular Age-Related Macular Degeneration: A Phase 3 Randomized Clinical Trial. JAMA Ophthalmol. 2023 Jul 1;141(7):668-676. doi: 10.1001/jamaophthalmol.2023.2260. PMID 37289448

RESULTS

PARTICIPANT FLOW:
Groups:
- SB15 (Proposed Aflibercept Biosimilar): Subjects who were randomized at Week 0 to receive SB15 (Aflibercept) every 4 weeks for the first 3 months (i.e., at Weeks 0, 4, and 8), followed by once every 8 weeks until Week 32.
  After re-randomization at Week 32, all the subjects continued to receive SB15 once every 8 weeks in transition period (Week 32 to Week 48).
- Eylea (Aflibercept): Subjects who were randomized at Week 0 to receive Eylea (Aflibercept) every 4 weeks for the first 3 months (i.e., at Weeks 0, 4, and 8), followed by once every 8 weeks until Week 32.
  After re-randomization at Week 32, subjects were transitioned to SB15 or Eylea 2mg (0.05 mL) once every 8 weeks in transition period (Week 32 to Week 48).
- Eylea (Aflibercept) to SB15: Subjects who were randomized at Week 0 to receive Eylea (Aflibercept) in the Main Period, and after re-randomization at Week 32, transitioned to receive SB15 (Aflibercept) once every 8 weeks in transition period (Week 32 to Week 48).
- Eylea (Aflibercept) to Eylea: Subjects who were randomized at Week 0 to receive Eylea (Aflibercept) in the Main Period, and after re-randomization at Week 32, continued to receive Eylea once every 8 weeks in transition period (Week 32 to Week 48).
Period: Main Period
Arm/Group | SB15 (Proposed Aflibercept Biosimilar) | Eylea (Aflibercept) | Eylea (Aflibercept) to SB15 | Eylea (Aflibercept) to Eylea
Started | 224 | 225 | 0 | 0
Completed | 219 | 219 | 0 | 0
Not Completed | 5 | 6 | 0 | 0
Period: Transition Period
Arm/Group | SB15 (Proposed Aflibercept Biosimilar) | Eylea (Aflibercept) | Eylea (Aflibercept) to SB15 | Eylea (Aflibercept) to Eylea
Started | 219 | 0 | 111 | 108
Completed | 215 | 0 | 109 | 101
Not Completed | 4 | 0 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Eylea (Aflibercept): Subjects randomized into Eylea group will receive Eylea 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
  At Week 32, subjects in Eylea group will re-randomized into SB15 or Eylea group. After re-randomization, subjects transited to SB15 group will receive SB15 2 mg (0.05 mL) once every 8 weeks until Week 48 and subjects remaining in Eylea group will continue to receive Eylea 2 mg (0.05 mL) once every 8 weeks until Week 48.
  SB15 (Proposed aflibercept biosimilar): Subjects randomized into SB15 group will receive SB15 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48. Starting at Week 32, subjects transited from Eylea to SB15 will receive SB15 2 mg (0.05 mL) via intravitreal injection every 8 weeks.
  Eylea (Aflibercept): Subjects randomized into Eylea group will receive Eylea 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
- Total: Total of all reporting groups
Arm/Group | SB15 (Proposed Aflibercept Biosimilar) | Eylea (Aflibercept) | Total
Number analyzed (Participants) | 224 | 225 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 23 | 56
  >=65 years | 191 | 202 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (8.05) | 74.3 (8.09) | 74.0 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 132 | 250
  Male | 106 | 93 | 199
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 51 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 170 | 172 | 342
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: The VA was assessed using original series ETDRS charts or 2702 series number charts.
Time Frame: Baseline and Week 8
Population: Primary outcome was analyzed on 448 subjects who were randomised at Week 0 in a 1:1 ratio to either SB15 or Eylea. Among 449 randomised subjects at Week 0, one subject in Eylea group did not receive IP during the study and was excluded from the analysis as pre-specified in analysis plan.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | SB15 (Proposed Aflibercept Biosimilar) | Eylea (Aflibercept)
Number analyzed (Participants) | 224 | 224
letters | 6.7 (0.56) | 6.6 (0.57)

ADVERSE EVENTS:
Time Frame: Overall Period (56 weeks)
Description: Safety analysis was performed on subjects who received at least one IP during the study period.
  Among 224 and 225 subjects initially randomised to SB15 and Eylea group, each of 224 and 224 subjects received the IP on Day 1.
  Safety analysis after Week 32 was performed on subjects who received at least one IP after re-randomisation.
  Among 111 and 108 subjects re-randomised to "Eylea to SB15" and "Eylea to Eylea" group, each of 111 and 104 subjects received at least one IP after Week 32.
Arm/Group | SB15 (Proposed Aflibercept Biosimilar) | Eylea (Aflibercept) | Eylea (Aflibercept) to SB15 | Eylea (Aflibercept) to Eylea
All-Cause Mortality (participants affected / at risk) | 1/224 | 2/224 | 0/111 | 1/104
Serious Adverse Events (participants affected / at risk) | 22/224 | 27/224 | 9/111 | 13/104
Other Adverse Events (participants affected / at risk) | 33/224 | 23/224 | 15/111 | 7/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB15 (Proposed Aflibercept Biosimilar) (N=224) | Eylea (Aflibercept) (N=224) | Eylea (Aflibercept) to SB15 (N=111) | Eylea (Aflibercept) to Eylea (N=104)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 1 | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Disease progression (General disorders) | 2 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Device placement issue (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ovarian clear cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB15 (Proposed Aflibercept Biosimilar) (N=224) | Eylea (Aflibercept) (N=224) | Eylea (Aflibercept) to SB15 (N=111) | Eylea (Aflibercept) to Eylea (N=104)
Neovascular age-related macular degeneration (Eye disorders) | 18 | 14 | 10 | 4
Visual acuity reduced (Eye disorders) | 15 | 11 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04450329/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04450329/SAP_001.pdf